CLINICAL TRIAL: NCT06185634
Title: Impact of Pasta Consumption Timing on Multiple Health Outcomes
Brief Title: Impact of the Timing of Pasta Consumption on Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Francesco Sofi, Professor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PASTA-TIMING
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Normal Weight
Keywords: Sleep quality; Anthropometric parameters; Mealtiming; Pasta; Cardiovascular risk; Gut microbiota
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The experimental study will be a randomised controlled trial and will involve 2 phases of nutritional intervention.
Masking Description: In this study it will not be possible to blind the experimenters and participants. Blinding will be impossible for the experimenters, as they will provide the food plan with the dietary intervention. Blinding will also not be possible for the participants, who will have to eat pasta only at dinner for 3 months and only at lunch for the same period of time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group starting with the dietary intervention of eating pasta at dinner for 3 months.
  Interventions: Other: Dietary intervention - Pasta at dinner; Other: Dietary intervention - Pasta at lunch
- Group 2 (Experimental): Group starting with the dietary intervention of eating pasta at lunch for 3 months.
  Interventions: Other: Dietary intervention - Pasta at dinner; Other: Dietary intervention - Pasta at lunch

INTERVENTIONS:
Other: Dietary intervention - Pasta at dinner — The "pasta at dinner" nutritional intervention will consist, as the name suggests, in eating pasta at dinner for 3 months. The dietary intervention will consist of a normo-caloric diet, defined on the basis of the individual basal metabolic rate measured by indirect calorimetry and on the calculation of the participant's calorie intake extrapolated from a 3-day food diary. The diet will be of the Mediterranean type with 30% of energy coming from fats, 15-20% from proteins and the remaining 50-55% from carbohydrates (mainly complexes). Calorie intake will be distributed as follows: 20% calories at breakfast, 5% calories in the mid-morning snack, 40% calories at lunch, 5% calories in the mid-afternoon snack, 30% calories at dinner.
Other: Dietary intervention - Pasta at lunch — The "pasta at lunch" nutritional intervention will consist, as the name suggests, in eating pasta at lunch for 3 months. The dietary intervention will consist of a normo-caloric diet, defined on the basis of the individual basal metabolic rate measured by indirect calorimetry and on the calculation of the participant's calorie intake extrapolated from a 3-day food diary. The diet will be of the Mediterranean type with 30% of energy coming from fats, 15-20% from proteins and the remaining 50-55% from carbohydrates (mainly complexes). Calorie intake will be distributed as follows: 20% calories at breakfast, 5% calories in the mid-morning snack, 40% calories at lunch, 5% calories in the mid-afternoon snack, 30% calories at dinner.

SUMMARY:
To date, the optimal timing for pasta consumption remains uncertain. Based on recent evidence in the field of chrono-nutrition, it is speculated that eating pasta at dinner may have a negative impact on cardio-metabolic health. Carbohydrate intake during a period of minimal glucose tolerance could potentially alter the glycaemic profile and increase the risk of overweight and obesity. Conversely, other studies indicate that consuming carbohydrates at dinner may enhance sleep efficiency and quality. Thus, the aim of this study is, for the first time, to evaluate whether there are discernible differences between consuming pasta at lunch or dinner for the human health.

DETAILED DESCRIPTION:
Background:

Pasta plays an indisputable role in the Mediterranean diet pyramid. Indeed, it is an excellent source of carbohydrates that can be part of a varied, balanced, and healthy diet. Despite this, more and more people are avoiding it because they consider it too caloric and associate it with weight gain, especially if eaten in the evening.

While it is known with certainty that the consumption of pasta, in the right quantities, is associated with positive health effects, there is limited information on the optimal time to consume it. The most common hypothesis is that it is better to consume it at lunch, as metabolism undergoes a physiological and progressive reduction as the evening approaches. Furthermore, recent findings in the field of chrono-nutrition have highlighted that glucose tolerance is high during the day and minimal during the night, suggesting that consuming a high amount of carbohydrates in the evening may predispose to weight gain and a worsened cardio-metabolic profile. On the other hand, according to some studies, consuming carbohydrates in the evening may ensure good sleep quality, as they are an excellent source of tryptophan, an amino acid that promotes serotonin production, also known as the sleep hormone.

Recently, some studies on animal models have suggested that the timing of carbohydrate consumption could also impact the composition and functionality of the gut microbiota. For example, it has been observed that the production of short-chain fatty acids (SCFA) fluctuates throughout the day under the control of the host's circadian rhythms. Considering that SCFA are produced from carbohydrates and are fundamental regulators for many metabolic processes, it could be extremely interesting to explore the relationship between "when carbohydrates are consumed" and microbial functionality.

In conclusion, to date, studies that have evaluated the timing of carbohydrate consumption are limited and rely on physiological and chrono-biological assumptions rather than experimental evidence. Consequently, it is not known whether consuming pasta at lunch or dinner, in the right quantities, may have effects on human weight and health.

Objective of the study:

The aim of this study is to assess, for the first time, whether there is a difference between consuming pasta at lunch or dinner in terms of sleep quality, anthropometric parameters, cardiovascular risk factors, composition and functionality of the gut microbiota in a sample of normal-weight subjects. Additionally, individual chronotype will be taken into consideration, a construct indicating when a subject is most active during the day, as recent studies have highlighted its impact on dietary habits, especially in terms of "meal timing," and human health.

ELIGIBILITY:
Inclusion Criteria:

* normal weight condition (BMI=18.5-24.9 kg/m2)
* age between 18 and 65 years
* willing to give informed consent

Exclusion Criteria:

* subjects who were involved in night work, planned long-distance jet travel during the study period, had irregular sleeping schedules or were taking any drugs known to affect sleep or metabolism
* presence of current chronic illness or unstable condition (e.g., cardiovascular disease, chronic liver disease, inflammatory bowel disease)
* current or recent (past 2 months) use of antibiotics or probiotics
* pregnancy or intention to become pregnant in the next 12 months
* breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-11-13 (Estimated); Study Completion 2025-11-13 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | 7 months
  The assessment of sleep quality will be done by actigraphy and the following parameters will be evaluated: sleep onset time, end of sleep time, waking after sleep onset, total sleep time, sleep efficiency, number of awakenings, duration of awakenings, movement index, activity index and sleep regularity index.This assessment will be carried out at the beginning and end of each of the two intervention phases.

SECONDARY OUTCOMES:
Weight change | 7 months
  Measurement of body weight change in kg at the beginning and end of each of the two intervention phases.
Body mass index (BMI) changes | 7 months
  Measurement of BMI change at the beginning and end of each of the two intervention phases. Weight and height will be combined to report BMI in kg/m^2
Fat mass changes | 7 months
  Measurement of fat mass change at the beginning and end of each of the two intervention phases. Percentage of fat mass will be assessed using the Akern bioelectrical impedance analyser (model SE 101).
Basal Metabolic Rate | 7 months
  Measurement of basale metabolic rate change at the beginning and end of each of the two intervention phases. The basal metabolism will be defined by indirect calorimetry.
Fasting Blood Glucose changes | 7 months
  Measurement of blood glucose concentration change in mg/dL at the beginning and end of each of the two intervention phases.
Glycated Haemoglobin (HbA1c) changes | 7 months
  Measurement of glycated haemoglobin (HbA1c) change in mmol/mol at the beginning and end of each of the two intervention phases.
Total cholesterol changes | 7 months
  Measurement of total cholesterol change in mg/dL at the beginning and end of each of the two intervention phases.
LDL-cholesterol changes | 7 months
  Measurement of LDL cholesterol change in mg/dL at the beginning and end of each of the two intervention phases.
HDL-cholesterol changes | 7 months
  Measurement of HDL cholesterol change in mg/dL at the beginning and end of each of the two intervention phases.
Triglycerides changes | 7 months
  Measurement of triglycerides change in mg/dL at the beginning and end of each of the two intervention phases.
Homocysteine changes | 7 months
  Measurement of homocysteine change in micromoli/L at the beginning and end of each of the two intervention phases.
Aspartate transaminase changes | 7 months
  Measurement of aspartate transaminase change in U/l at the beginning and end of each of the two intervention phases.
Alanine transaminase changes | 7 months
  Measurement of alanine transaminase change in U/l at the beginning and end of each of the two intervention phases.
Gamma-glutamyl transferase changes | 7 months
  Measurement of gamma-glutamyl transferase change in U/l at the beginning and end of each of the two intervention phases.
Urea changes | 7 months
  Measurement of urea change in mg/dL at the beginning and end of each of the two intervention phases.
Creatinine changes | 7 months
  Measurement of creatinine change in mg/dL at the beginning and end of each of the two intervention phases.
Uric acid changes | 7 months
  Measurement of uric acid change in mg/dL at the beginning and end of each of the two intervention phases.
Gut microbiota changes | 7 months
  Measurement of gut microbiota profile change at the beginning and end of each of the two intervention phases. Each subject will be asked for a stool sample at the beginning and at the end of each intervention phases in order to analyse the composition of the gut microbiota and short-chain fatty acids production.
Individual circadian rhythms | 7 months
  Circadian rhythms and the individual chronotype will be analysed for each participant through the Dim Light Melatonin Onset (DMLO) at the beginning and end of each of the two intervention phases. For this purpose, the NovoLytiX ELISA kit for Direct Melatonin on Saliva (EK-DSM) will be used.
TBARS changes | 7 months
  Measurement of TBARS changes at the beginning and end of each of the two intervention phases.
ROS changes | 7 months
  Measurement of ROS changes at the beginning and end of each of the two intervention phases.
Leptin changes | 7 months
  Measurement of leptin changes at the beginning and end of each of the two intervention phases.
Ghrelin changes | 7 months
  Measurement of ghrelin changes at the beginning and end of each of the two intervention phases.
Insulin changes | 7 months
  Measurement of insulin changes at the beginning and end of each of the two intervention phases.
IL-6 changes | 7 months
  Measurement of IL-6 changes at the beginning and end of each of the two intervention phases.
C-Peptide YY | 7 months
  Measurement of C-Peptide YY changes at the beginning and end of each of the two intervention phases.

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Clinical Nutrition, University Hospital of Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang M, Lo K, Li J, Allison M, Wu WC, Liu S. Pasta meal intake in relation to risks of type 2 diabetes and atherosclerotic cardiovascular disease in postmenopausal women : findings from the Women's Health Initiative. BMJ Nutr Prev Health. 2021 Apr 30;4(1):195-205. doi: 10.1136/bmjnph-2020-000198. eCollection 2021. PMID 34308127
- [Background] Henry CJ, Kaur B, Quek RYC. Chrononutrition in the management of diabetes. Nutr Diabetes. 2020 Feb 19;10(1):6. doi: 10.1038/s41387-020-0109-6. PMID 32075959
- [Background] St-Onge MP, Mikic A, Pietrolungo CE. Effects of Diet on Sleep Quality. Adv Nutr. 2016 Sep 15;7(5):938-49. doi: 10.3945/an.116.012336. Print 2016 Sep. PMID 27633109
- [Background] Frazier K, Chang EB. Intersection of the Gut Microbiome and Circadian Rhythms in Metabolism. Trends Endocrinol Metab. 2020 Jan;31(1):25-36. doi: 10.1016/j.tem.2019.08.013. Epub 2019 Oct 31. PMID 31677970
- [Background] la Fleur SE, Kalsbeek A, Wortel J, Fekkes ML, Buijs RM. A daily rhythm in glucose tolerance: a role for the suprachiasmatic nucleus. Diabetes. 2001 Jun;50(6):1237-43. doi: 10.2337/diabetes.50.6.1237. PMID 11375322
- [Background] Afaghi A, O'Connor H, Chow CM. High-glycemic-index carbohydrate meals shorten sleep onset. Am J Clin Nutr. 2007 Feb;85(2):426-30. doi: 10.1093/ajcn/85.2.426. PMID 17284739
- [Background] Thaiss CA, Levy M, Korem T, Dohnalova L, Shapiro H, Jaitin DA, David E, Winter DR, Gury-BenAri M, Tatirovsky E, Tuganbaev T, Federici S, Zmora N, Zeevi D, Dori-Bachash M, Pevsner-Fischer M, Kartvelishvily E, Brandis A, Harmelin A, Shibolet O, Halpern Z, Honda K, Amit I, Segal E, Elinav E. Microbiota Diurnal Rhythmicity Programs Host Transcriptome Oscillations. Cell. 2016 Dec 1;167(6):1495-1510.e12. doi: 10.1016/j.cell.2016.11.003. PMID 27912059
- [Background] Zhao M, Tuo H, Wang S, Zhao L. The Effects of Dietary Nutrition on Sleep and Sleep Disorders. Mediators Inflamm. 2020 Jun 25;2020:3142874. doi: 10.1155/2020/3142874. eCollection 2020. PMID 32684833
- [Background] Gerard C, Vidal H. Impact of Gut Microbiota on Host Glycemic Control. Front Endocrinol (Lausanne). 2019 Jan 30;10:29. doi: 10.3389/fendo.2019.00029. eCollection 2019. PMID 30761090
- [Background] Lotti S, Pagliai G, Colombini B, Sofi F, Dinu M. Chronotype Differences in Energy Intake, Cardiometabolic Risk Parameters, Cancer, and Depression: A Systematic Review with Meta-Analysis of Observational Studies. Adv Nutr. 2022 Feb 1;13(1):269-281. doi: 10.1093/advances/nmab115. PMID 34549270
- [Derived] Lotti S, Dinu M, Napoletano A, Pagliai G, Asensi MT, Giangrandi I, Cesari F, Becatti M, Amedei A, Fiorillo C, Marcucci R, Colombini B, Sofi F. The impact of the timing of pasta intake on sleep quality and health outcomes: a protocol for a randomized controlled trial. Trials. 2025 May 8;26(1):150. doi: 10.1186/s13063-025-08859-x. PMID 40340858